CLINICAL TRIAL: NCT06685484
Title: A Study on the Feasibility of Modified Mindfulness Training Program (MMTP) to Address Antenatal Depression and Perceived Stress Among Pregnant Women Exhibiting Male Child Preference
Brief Title: Feasibility of Modified Mindfulness Training on Antenatal Depression and Perceived Stress in Pregnant Women With Male Child Preference
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khyber Medical University Peshawar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KMU/DIR/CTU/2024/009
Record Dates: First submitted 2024-11-05; First posted 2024-11-12 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Antenatal Depression
Keywords: Mindfulness training; Antenatal depression; Male Child preference; Perceived Stress

STUDY DESIGN:
Intervention Model Description: A feasibility trial using the ADAPT-ITT framework will randomly assign participants to two groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Receives Modified Mindfulness Training Program (MMTP), adapted to address cultural stressors and reduce antenatal depression.
  Interventions: Behavioral: Modified Mindfulness Training Program (MMTP)
- Control Group (No Intervention): Receives standard antenatal care without mindfulness intervention.

INTERVENTIONS:
Behavioral: Modified Mindfulness Training Program (MMTP) — The intervention, designed as a Modified Mindfulness Training Program (MMTP), aims to reduce antenatal depression and perceived stress among pregnant women, especially those with a preference for a male child. This program is adapted to address culturally specific stressors relevant to these women, promoting mental health and resilience during pregnancy.
  The intervention is based on Nola Pender's Health Promotion Model and structured using the ADAPT-ITT framework, which includes Assessment, Decision, Adaptation, Production, Topical Experts, Integration, Training, and Testing phases. This phased approach ensures cultural relevance and feasibility within the target population of pregnant women in Pakistan.
  Duration and Frequency: The intervention consists of six weekly sessions, each lasting two hours, held in a serene, controlled environment within a seminar room at Sindh Govt. Qatar Hospital, Karachi.
  Arms: Intervention Group

SUMMARY:
This study will assess the feasibility of a modified mindfulness training intervention aimed at reducing antenatal depression and perceived stress in pregnant women with male child preference. The findings aim to support mental health interventions in maternity care.

DETAILED DESCRIPTION:
Utilizing the ADAPT-ITT framework, this study will tailor mindfulness-based interventions to address unique cultural stressors, particularly those affecting maternal mental health due to male child preference.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in the first and second trimester
* Score ≥10 on the Edinburgh Postnatal Depression Scale (EPDS)

Exclusion Criteria:

* Psychiatric illness history, use of psychiatric medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-04-23 (Actual)

PRIMARY OUTCOMES:
Reduction in Antenatal Depression | Baseline assessment, immediately post-intervention (six weeks), and one-month follow-up.
  This outcome specifically measures changes in antenatal depression levels among pregnant women with male child preference. Depression will be assessed using the Edinburgh Postnatal Depression Scale (EPDS), with scores taken at baseline, immediately post-intervention, and at the one-month follow-up. A reduction in EPDS scores from baseline to follow-up indicates improvement in mental health.
Reduction in Perceived Stress | Immediately post-intervention (after six weeks)
  This outcome focuses on changes in perceived stress levels using the Perceived Stress Scale (PSS-10). Scores will be taken at baseline, post-intervention, and one-month follow-up to measure the effectiveness of the Modified Mindfulness Training Program (MMTP) on stress reduction.
Participant Satisfaction with the Modified Mindfulness Training Program | Immediately post-intervention (after six weeks)
  This outcome measures participant satisfaction levels with the Modified Mindfulness Training Program intervention, gauging ease of use, cultural appropriateness, and overall program relevance. Data will be gathered using a post-intervention feedback survey with Likert-scale responses.
Acceptability of the Modified Mindfulness Training Program in a Clinical Setting | Immediately post-intervention (after six weeks)
  This outcome evaluates the acceptability of the Modified Mindfulness Training Program intervention in a clinical setting, using qualitative data from open-ended interviews. The qualitative feedback will indicate cultural appropriateness and feasibility of implementation.
Follow-Up Effects on Coping Skills | One-month follow-up after intervention completion
  This outcome assesses sustained improvements in coping skills for managing antenatal stress post-intervention, measured through scores on the PSS-10 at one-month follow-up.
Follow-Up Effects on Resilience | One-month follow-up after intervention completion
  This outcome focuses on the resilience of participants in managing antenatal depression, measured through EPDS scores and supported by qualitative feedback at one-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Badil, Principal Investigator — Institute of Nursing Sciences, Khyber Medical University Peshawar; Dr Najma Naz, PhD, Principal Investigator — Institute of Nursing, Khyber Medical University Peshawar; Dr Khalid Rahman, PhD, Principal Investigator — Institute of Public Health and Social Science, Khyber Medical University Peshawar
Locations (1):
- Qatar Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
The IPD sharing plan includes de-identified data for the primary and secondary outcomes, specifically related to antenatal depression and perceived stress scores (PSS-10 and EPDS) before and after the intervention, as well as demographic information that may influence outcomes (e.g., age, pregnancy stage, gender preference). The data will be shared to facilitate replication studies, meta-analyses, and further research on the Modified Mindfulness Training Program's effects on antenatal mental health.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available six months after the primary study publication and remain accessible for three years.
Access Criteria: Researchers can request access to IPD via a formal application process, which includes justification for use, research objectives, and adherence to data privacy agreements. Access will be granted to qualified researchers following review and approval by the data-sharing committee.

REFERENCES:
- [Background] Ayano G, Tesfaw G, Shumet S. Prevalence and determinants of antenatal depression in Ethiopia: A systematic review and meta-analysis. PLoS One. 2019 Feb 19;14(2):e0211764. doi: 10.1371/journal.pone.0211764. eCollection 2019. PMID 30779765
- [Background] Guo J, Zheng A, He J, Ai M, Gan Y, Zhang Q, Chen L, Liang S, Yu X, Kuang L. The prevalence of and factors associated with antenatal depression among all pregnant women first attending antenatal care: a cross-sectional study in a comprehensive teaching hospital. BMC Pregnancy Childbirth. 2021 Oct 26;21(1):713. doi: 10.1186/s12884-021-04090-z. PMID 34702205
- [Background] Yin X, Sun N, Jiang N, Xu X, Gan Y, Zhang J, Qiu L, Yang C, Shi X, Chang J, Gong Y. Prevalence and associated factors of antenatal depression: Systematic reviews and meta-analyses. Clin Psychol Rev. 2021 Feb;83:101932. doi: 10.1016/j.cpr.2020.101932. Epub 2020 Oct 25. PMID 33176244
- [Background] Sikander S, Ahmad I, Bates LM, Gallis J, Hagaman A, O'Donnell K, Turner EL, Zaidi A, Rahman A, Maselko J. Cohort Profile: Perinatal depression and child socioemotional development ; the Bachpan cohort study from rural Pakistan. BMJ Open. 2019 May 5;9(5):e025644. doi: 10.1136/bmjopen-2018-025644. PMID 31061029
- [Background] Tesfaye Y, Agenagnew L. Antenatal Depression and Associated Factors among Pregnant Women Attending Antenatal Care Service in Kochi Health Center, Jimma Town, Ethiopia. J Pregnancy. 2021 Feb 8;2021:5047432. doi: 10.1155/2021/5047432. eCollection 2021. PMID 33628509